CLINICAL TRIAL: NCT06676891
Title: Expanded Access to RZ-001 in Combination with Valganciclovir in the Treatment of Subjects with Glioblastoma
Brief Title: Expanded Access Program for GBM Subjects
Status: Available | Type: Expanded Access
Sponsor: Rznomics, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RZ-001-201-EAP
Record Dates: First submitted 2024-10-27; First posted 2024-11-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: RZ-001 — Participants will receive a single intracerebral injection of RZ-001, Recombinant adenovirus harboring the modified ribozyme construct with HSV-tk as a therapeutic transgene

SUMMARY:
This small-size patient population expanded access program is to provide access to investigational product RZ-001 for up to around 4 patients with human telomerase reverse transcriptase(hTERT)-positive Glioblastoma (GBM) who are not eligible to participate in the RZ-001-201 clinical study or in any other study involving the use of RZ-001

DETAILED DESCRIPTION:
This expanded access protocol provides expanded access to RZ-001 to patients with glioblastoma. After provision of written informed consent, subjects will be evaluated for eligibility during the Screening period, a period of 28 days prior to the RZ-001 administration on Day 1. Subjects will then undergo treatment, 8 weeks of follow-up, and bimonthly or quarterly (after 6 months from RZ-001 administration) survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females legally considered to be adults in the country in which they are participating in the study.
2. Histologically-confirmed Grade 4 astrocytoma, GBM, per The 2021 WHO Classification of central nervous system (CNS) Tumors.
3. Recurrent GBM with radiographic evidence of the PD (progressive disease) which contains measurable disease (≥ 1 cm bidirectional diameters) by contrast-enhancement on MRI, as defined by the mRANO (modified Response Assessment in Neuro-Oncology) criteria. Only localized unifocal or multifocal recurrence is allowed, while other type of recurrences such as intraventricular, diffuse recurrence are not allowed.

Exclusion Criteria:

1. Diagnosis of other malignant tumors within 5 years prior to RZ-001 administration.
2. Have received chemotherapy within 4 weeks, and/or immunomodulatory therapy, immunotherapy, antibody therapy, gene vector therapy, vaccine therapy, and/or matrix metalloprotease inhibitor(s) within 3 months from Screening.
3. Have received radiotherapy within 12 weeks from Screening.
4. Have extracranial metastases of the tumor cells.
5. The subject is eligible for participation in any ongoing clinical study with RZ-001, or has already received RZ-001 in the past.
6. The subject is being transferred from an ongoing clinical study for which they are still eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States